CLINICAL TRIAL: NCT00715871
Title: Phase II Study to Measure Effectiveness and to Monitor Side Effects of Smoke-Break Nicotine Delivery Device
Brief Title: Clinical Study of Smoke-Break Liquid Cigarettes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Smoke-Break, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB07211
Record Dates: First submitted 2008-07-08; First posted 2008-07-15 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Smoking
Keywords: smoking; smoke cessation; stop smoking; quit smoking; nicotine replacement therapy; Smoke Break; liquid cigarette; liquid nicotine cigarette
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Smokers (Experimental): Active smokers who used the Smoke-Break nicotine delivery device in an attempt to quit smoking cigarettes.
  Interventions: Drug: Nicotine; Device: Smoke-Break nicotine delivery device

INTERVENTIONS:
Drug: Nicotine — Subjects received an amount of "liquid nicotine cigarettes" (containing 1.5mg of nicotine each) based on the amount of nicotine the subjects had been receiving from cigarettes. The number of "liquid nicotine cigarettes" received by each subject was reviewed, and adjusted (if necessary), every two weeks for the duration of the 12-week study.
  Other Names: Smoke-Break, liquid cigarette, liquid nicotine cigarette
Device: Smoke-Break nicotine delivery device — The Smoke-Break nicotine delivery device is a "liquid nicotine cigarette" designed to mimic the act of smoking. It is an NRT (nicotine replacement therapy) similar in concept to the nicotine patch, gum, and lozenge, except the nicotine is delivered in a way designed to duplicate the cigarette smoking experience. The Smoke-Break nicotine delivery device is non-invasive.
  Other Names: Smoke-Break, liquid cigarette, liquid nicotine cigarette

SUMMARY:
The purpose of this study is to determine whether the Smoke-Break nicotine delivery device can help smokers quit smoking, while avoiding many of the side effects associated with other smoking cessation products.

DETAILED DESCRIPTION:
The study has been completed and published. The published study manuscript can be found here: http://www.biomedcentral.com/1471-2458/10/155

ELIGIBILITY:
Inclusion Criteria:

* Volunteer is at least 18 years of age.
* Volunteer currently smokes cigarettes, cigars or other forms of tobacco products for at least one year.
* Volunteer wants to quit smoking.
* Volunteer will be fully informed as to the nature of the study.
* Volunteer will have no known allergy to any product ingredients as listed in the informed consent.
* Volunteer agrees to a confidential pretest questionnaire and periodic monitoring as to the effectiveness of the smoking cessation regimen.
* Volunteers are not currently using another nicotine replacement therapy.
* Volunteer will agree to use birth control measures while on the study.

Exclusion Criteria:

* Volunteer has a known allergy or hypersensitivity to nicotine or other related ingredients as outlined in the informed consent.
* Volunteer does not desire to quit smoking.
* Volunteer is using another nicotine replacement therapy.
* Volunteer is pregnant or breast-feeding.
* Volunteer has a history of heart disease or advanced diabetes.
* Volunteer indicates on the application that they smoke ten (10) or fewer cigarettes per day.
* Volunteer is using a daily prescription medicine for depression or asthma.
* Volunteer is using a non-nicotine smoke cessation drug, such as Zyban or Chantix.
* Volunteer is an employee of Smoke-Break Inc., or is personally known to an employee of Smoke-Break Inc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Smoke cessation | 12 weeks

SECONDARY OUTCOMES:
Side effects | 0-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Geimer, MD, Principal Investigator — Smoke-Break, Inc.
Locations (1):
- Tommy G. Thompson Youth Center, West Allis, Wisconsin, United States

REFERENCES:
- [Derived] Geimer N, Olson CE, Baumgarten D, Kepner JL, Mahoney MC. Use of a liquid nicotine delivery product to promote smoking cessation. BMC Public Health. 2010 Mar 24;10:155. doi: 10.1186/1471-2458-10-155. PMID 20334673